CLINICAL TRIAL: NCT01307891
Title: An Open Label, Randomized, Phase II Trial of Abraxane (Paclitaxel Albumin-Bound Particles for Injectable Suspension), With or Without Tigatuzumab (a Humanized Monoclonal Antibody Targeting Death Receptor 5) in Patients With Metastatic, Triple Negative (ER, PR, and HER-2 Negative) Breast Cancer
Brief Title: Abraxane With or Without Tigatuzumab in Patients With Metastatic, Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Daiichi Sankyo UK Ltd. (Other); Triple Negative Breast Cancer Foundation (Unknown)
Responsible Party: Principal Investigator, Andres Forero, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F101004001 (UAB1028); TBCRC 019 (Other: The Translational Breast Cancer Research Consortium)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Stage IV Breast Cancer; Metastatic Breast Cancer
Keywords: Triple negative breast cancer (TNBC); Metastatic breast cancer; Tigatuzumab (CS-1008); Abraxane (ABI-007); HER-2-neu negative; ER negative, PR negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; tigatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abraxane + Tigatuzumab (Experimental): Patients will receive Abraxane at 100 mg/m2 X 3 doses on Days 1, 8, and 15 at 28-day intervals and tigatuzumab to be administered as a 10 mg/kg loading dose followed by 5 mg/kg for the first cycle and then every other week on Days 1 and 15 for subsequent cycles. Patients will be evaluated for response every 8 weeks. Patients with disease progression will be taken off the study.
  Interventions: Drug: Abraxane + Tigatuzumab
- Abraxane alone (Experimental): Patients will receive Abraxane at 100 mg/m2 weekly X 3 doses on Days 1, 8, and 15 at 28-day intervals. Patients will have the option to crossover to the combination arm based upon the pre-clinical data.
  Interventions: Drug: Abraxane alone

INTERVENTIONS:
Drug: Abraxane alone — 100 mg/m2 weekly X 3 doses (Days 1, 8, 15) at 28-day intervals until disease progression or unacceptable toxicity. Abraxane will be administered on an outpatient basis by an IV infusion over 30 minutes. Patients will be evaluated for response every 2 cycles (every 8 weeks).
  Other Names: Abraxane, also ABI-007
  Arms: Abraxane alone
Drug: Abraxane + Tigatuzumab — Tigatuzumab will be administered as a loading dose of 10 mg/kg on Day 1, then 5 mg/kg on Day 15 and then every other week on Days 1 and 15 of subsequent cycles. It will be given as an IV infusion over 60 minutes or less. No dose reductions will be allowed. Tigatuzumab will be administered in combination with the Abraxane according to the intervention described for it.
  Other Names: Tigatuzumab, CS-1008
  Arms: Abraxane + Tigatuzumab

SUMMARY:
Breast cancer is the most commonly diagnosed cancer and the second leading cause of cancer deaths in American women. Metastatic disease including metastatic breast cancer unfortunately remains incurable. One reason is due to the inability to develop specific therapies for specific cancer subsets.

The use of modern genomic techniques has significantly enhanced our recent understanding of breast cancer biology. Five distinct breast cancer subsets have been recognized, one of which is basal-like breast cancer. Basal-like breast cancer is typically estrogen receptor (ER) negative, progesterone receptor (PR) negative and human epidermal growth factor receptor 2 (HER-2-Neu) negative. This is referred to as triple negative breast cancer or TBNC. TBNC represents a significant proportion of breast cancer patients (10-20%) and has a poor prognosis with no targeted approach to therapy as of yet.

Tigatuzumab is a humanized monoclonal antibody targeting a death receptor on the breast cancer cells. Previous studies have shown that combining antibodies with selected chemotherapy agents have induced tumor cell death. The hypothesis of this study is to use tigatuzumab and combine it with Abraxane to serve as a targeting agent in metastatic TBNC patients.

DETAILED DESCRIPTION:
The study is an open-label randomized, multi-institutional, phase II clinical trial of Abraxane in combination with tigatuzumab or Abraxane as a single agent in patients with TNBC. Randomization (2:1) will be made from these two categories: TBNC patients with no prior chemotherapy for metastatic disease or TBNC patients with prior taxane (except Abraxane) therapy for metastatic disease. Patients randomized to Abraxane alone may be allowed to cross over to the combination of Abraxane + tigatuzumab if there is disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented Stage IV breast cancer. If blocks (paraffin-embedded tissue) from original diagnosis are available, they will be obtained to confirm the diagnosis and for correlative studies. Fifteen slides can be obtained from the block if the block is not available to be sent or released.
* Tumor must be HER-2-neu negative (defined as 0 or 1+ staining by immunohistochemistry or gene amplification ratio less than or equal to 2.0, by fluorescent in situ hybridization - FISH), estrogen and progesterone receptors negative (<10%).
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded)
* Biopsy of a metastatic lesion is not required for protocol entry but all patients with reasonably accessible lesions (chest wall, breast, skin, subcutaneous, superficial lymph nodes, bones and liver metastases) must agree to biopsy.

  1. Biopsies may be done with local anesthesia or intravenous conscious sedation, according to standard institutional guidelines.
  2. If a biopsy requires general anesthesia, then it is only allowed if acquisition of tissue is necessary for clinical reasons and excess tissue that would otherwise have been discarded is then used for research purposes. If a biopsy requires general anesthesia, then a biopsy of that site for research purposes only, without a coexisting clinical indication is not allowed on this protocol.
  3. Patients with reasonably accessible lesions as described above, who will not agree with the biopsy, will not be enrolled in the trial.
  4. Patients with NO reasonably accessible lesions as described above can be enrolled in the trial.

Prior Therapy:

* There is no restriction as to the number of prior regimens for metastatic disease as long as patients have adequate performance status. Patients with no prior chemotherapy for metastatic disease and patients who have received prior therapy with taxanes for metastatic disease (taxol or taxotere) are eligible. Stratification will be used for randomization of these two categories (no prior chemotherapy for metastatic disease or prior taxane therapy for metastatic disease).
* Chemotherapy treatment prior to enrollment must be discontinued for at least 3 weeks prior to study entry.
* Patients must have completed radiation therapy at least 7 days prior to beginning protocol treatment.
* Patients must have recovered from all reversible toxicities related to prior therapy before beginning protocol treatment, and may not have any pre- existing treatment-related toxicities in excess of grade 1. Patients must have < grade 2 pre-existing peripheral neuropathy.
* Patients may receive bisphosphonates; however, if used, bone lesions may not be used for progression or response.
* At least 18 years of age (19 in Alabama).
* Life expectancy of greater than 12 weeks.
* ECOG performance status < or equal to 2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count: > or equal to 1,500/mcL,
  * Hemoglobin: > or equal to 9 mg/dL,
  * Platelets: > or equal to 100,000/mcL,
  * Total bilirubin: < or equal to 1.5 X institutional upper limit of normal,
  * AST(SGOT)/ALT(SGPT): < or equal to 2.5 X institutional upper limit of normal without liver metastases, OR < or equal to 5 X institutional upper limit of normal if documented liver metastases,
  * Creatinine: < or equal to 2.0 mg/dL, OR calculated creatinine clearance greater than or equal to 50 mL/min (calculated by the Cockcroft and Gault method).
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women are eligible.
* Use of an effective means of contraception in subjects of child-bearing potential.
* Negative serum or urine beta-HCG pregnancy test at screening for patients with childbearing potential.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Prior use of Abraxane for metastatic disease or in the adjuvant setting.
* Metastatic lesions identifiable only by PET.
* Patients may not be receiving concurrent chemotherapy for treatment of metastatic disease.
* Active brain metastases: evidence of progression < or equal to 3 months after local therapy (patients should be asymptomatic and off corticosteroids and anticonvulsants for at least 3 months prior to study entry).
* Patients with brain metastases must have at least one site of measurable disease outside of the central nervous system.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, history of recent myocardial infarction, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated. These potential risks may also apply to other agents used in this study.
* A prior invasive malignant disease within five years except for skin cancer (squamous cell or basal cell carcinoma).
* Patients with known history of HIV or Hepatitis B because of potential for added toxicity from treatment regimen.
* Dementia or altered mental status that would prohibit the understanding of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Center Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong YT, Zhang LJ, Liu YC, Tang M, Lin JY, Chen XY, Chen YX, Yan Y, Zhang WD, Jin JM, Luan X. Neutrophils as potential therapeutic targets for breast cancer. Pharmacol Res. 2023 Dec;198:106996. doi: 10.1016/j.phrs.2023.106996. Epub 2023 Nov 14. PMID 37972723

RESULTS

PARTICIPANT FLOW:
Groups:
- Abraxane Alone: Patients will receive Abraxane at 100 mg/m2 weekly X 3 doses on Days 1, 8, and 15 at 28-day intervals. Abraxane will be administered on an outpatient basis by an IV infusion over 30 minutes. Patients will be evaluated for response every 2 cycles (every 8 weeks).
Period: Overall Study
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone
Started | 42 | 22
Completed | 39 | 21
Not Completed | 3 | 1
Not completed — Progressive Disease | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone | Total
Number analyzed (Participants) | 42 | 22 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 18 | 53
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 22 | 64
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 26 | 16 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 42 | 22 | 64

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Patient response rates will be measured by the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI. Responses include the following: Complete Response (CR) disappearance of all target lesions; Partial Response (PR) at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) best response from the start of treatment until disease progression.
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone
Number analyzed (Participants) | 39 | 21
percentage of patients | 28 [14.9 to 45.0] | 38 [18 to 61.1]

2. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Patients will be assessed throughout the study for Grade 4 or 5 toxicities utilizing the Common Toxicity Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone
Number analyzed (Participants) | 39 | 21
Participants | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Baseline through 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone
Number analyzed (Participants) | 39 | 21
months | 2.8 [1.9 to 3.6] | 3.8 [2.8 to 19.7]

ADVERSE EVENTS:
Time Frame: Baseline to 24 months
Groups:
- Abraxane + Tigatuzumab: Patients will receive Abraxane at 100 mg/m2 X 3 doses on Days 1, 8, and 15 at 28-day intervals and tigatuzumab to be administered as a 10 mg/kg loading dose followed by 5 mg/kg for the first cycle and then every other week on Days 1 and 15 for subsequent cycles. Patients will be evaluated for response every 8 weeks.
- Abraxane Alone: Patients will receive Abraxane at 100 mg/m2 weekly X 3 doses on Days 1, 8, and 15 at 28-day intervals. Patients will have the option to crossover to the combination arm based upon the pre-clinical data. Abraxane will be administered on an outpatient basis by an IV infusion over 30 minutes. Patients will be evaluated for response every 2 cycles (every 8 weeks).
Arm/Group | Abraxane + Tigatuzumab | Abraxane Alone
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/39 | 3/21
Other Adverse Events (participants affected / at risk) | 39/39 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abraxane + Tigatuzumab (N=39) | Abraxane Alone (N=21)
Fever (Infections and infestations) | 1 (39) | 1 (21)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Empyema associated with a permanent thoracic catheter (Infections and infestations) | 1 (1) | 0 (0)
Bilateral Pulmonary Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abraxane + Tigatuzumab (N=39) | Abraxane Alone (N=21)
Fatigue (General disorders) | 22 (22) | 11 (11)
Alopecia (General disorders) | 19 (19) | 11 (11)
Pheripheral Sensory Neuropathy (Nervous system disorders) | 17 (17) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 16 (16) | 9 (9)
Nausea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No